CLINICAL TRIAL: NCT03511846
Title: The Pain Biomarker Study: Changes in Circulating Pain Signalling Molecules with Activation of Pain Receptors
Brief Title: Pain Biomarker Study
Acronym: PBS
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Mark J Burish, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: HSC-MS-17-0763
Record Dates: First submitted 2018-04-17; First posted 2018-04-30 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Migraine; Cluster Headache; Trigeminal Autonomic Cephalgia; Hemicrania Continua; Paroxysmal Hemicrania; SUNCT; Short-Lasting Unilateral Neuralgiform Headache with Conjunctival Injection and Tearing
Keywords: Brain Freeze; Capsaicin
MeSH Terms: conditions — Migraine Disorders; Cluster Headache; Trigeminal Autonomic Cephalalgias; Paroxysmal Hemicrania; Lacerations | interventions — Capsaicin; Air

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: In the oxygen portion of the study, subjects and the outcomes assessors will be told that they will be receiving either medical air or oxygen.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (16):
- Oral capsaicin (Experimental)
  Interventions: Drug: Oral capsaicin
- Oral capsaicin and Medical Air (Sham Comparator)
  Interventions: Drug: Oral capsaicin; Other: Medical Air
- Oral Capsaicin and Low Flow Oxygen (Experimental)
  Interventions: Drug: Oral capsaicin; Drug: Low Flow Oxygen
- Oral capsaicin and High Flow Oxygen (Experimental)
  Interventions: Drug: Oral capsaicin; Drug: High Flow Oxygen
- Topical capsaicin (Experimental)
  Interventions: Drug: Topical capsaicin
- Topical capsaicin and Medical Air (Sham Comparator)
  Interventions: Drug: Topical capsaicin; Other: Medical Air
- Topical capsaicin and Low Flow Oxygen (Experimental)
  Interventions: Drug: Topical capsaicin; Drug: Low Flow Oxygen
- Topical capsaicin and High Flow Oxygen (Experimental)
  Interventions: Drug: Topical capsaicin; Drug: High Flow Oxygen
- Intranasal capsaicin (Experimental)
  Interventions: Drug: Intranasal capsaicin
- Intranasal capsaicin and Medical Air (Sham Comparator)
  Interventions: Drug: Intranasal capsaicin; Other: Medical Air
- Intranasal capsaicin and Low Flow Oxygen (Experimental)
  Interventions: Drug: Intranasal capsaicin; Drug: Low Flow Oxygen
- Intranasal capsaicin and High Flow Oxygen (Experimental)
  Interventions: Drug: Intranasal capsaicin; Drug: High Flow Oxygen
- Cold water irrigation (Experimental)
  Interventions: Other: Cold Water Irrigation
- Cold water irrigation and Medical Air (Sham Comparator)
  Interventions: Other: Cold Water Irrigation; Other: Medical Air
- Cold water irrigation and Low Flow Oxygen (Experimental)
  Interventions: Other: Cold Water Irrigation; Drug: Low Flow Oxygen
- Cold water irrigation and High Flow Oxygen (Experimental)
  Interventions: Other: Cold Water Irrigation; Drug: High Flow Oxygen

INTERVENTIONS:
Drug: Oral capsaicin — Subjects will drink a solution with capsaicin
  Arms: Oral Capsaicin and Low Flow Oxygen; Oral capsaicin; Oral capsaicin and High Flow Oxygen; Oral capsaicin and Medical Air
Drug: Topical capsaicin — Capsaicin cream will be applied to the skin of the forehead, cheek, or leg
  Arms: Topical capsaicin; Topical capsaicin and High Flow Oxygen; Topical capsaicin and Low Flow Oxygen; Topical capsaicin and Medical Air
Drug: Intranasal capsaicin — Capsaicin cream will be applied to the nostril
  Arms: Intranasal capsaicin; Intranasal capsaicin and High Flow Oxygen; Intranasal capsaicin and Low Flow Oxygen; Intranasal capsaicin and Medical Air
Other: Cold Water Irrigation — Subjects will be asked to drink up to 2000 ml of cold water or ice water (temperature 0-10 degrees Celsius) as fast as possible, either continuously or intermittently (i.e. 200-800 ml at a time)
  Arms: Cold water irrigation; Cold water irrigation and High Flow Oxygen; Cold water irrigation and Low Flow Oxygen; Cold water irrigation and Medical Air
Other: Medical Air — Subjects will be exposed to medical air
  Arms: Cold water irrigation and Medical Air; Intranasal capsaicin and Medical Air; Oral capsaicin and Medical Air; Topical capsaicin and Medical Air
Drug: Low Flow Oxygen — Subjects will be exposed to oxygen gas between 1-9 L/min
  Arms: Cold water irrigation and Low Flow Oxygen; Intranasal capsaicin and Low Flow Oxygen; Oral Capsaicin and Low Flow Oxygen; Topical capsaicin and Low Flow Oxygen
Drug: High Flow Oxygen — Subjects will be exposed to oxygen gas between 10-25 L/min
  Arms: Cold water irrigation and High Flow Oxygen; Intranasal capsaicin and High Flow Oxygen; Oral capsaicin and High Flow Oxygen; Topical capsaicin and High Flow Oxygen

SUMMARY:
This study investigates molecular and physical biomarkers of headaches in order to better understand mechanisms of these diseases.

There are 3 main parts:

1. Use of capsaicin (active ingredient in hot chili peppers) to trigger release of calcitonin gene related peptide - the hypothesis is that this will be different in headache subjects compared to controls (and if so might be used to predict how these patients will respond to certain medications that modulate calcitonin gene-related peptide). Subjects will be given capsaicin as a cream applied to the forehead or the inner nostril, or a hot sauce that is ingested.
2. Use of capsaicin to trigger eye watering - the hypothesis is that oxygen gas will slow down the amount of eye watering. Cluster headache patients respond very powerfully to oxygen gas but to very little else. The mechanism for oxygen is unknown but in rodents there is data that it works on the parasympathetic / lacrimal gland system. This study translates rodent data into humans in a non-invasive way to confirm the mechanism of this very effective treatment.
3. Use of ice water to trigger headaches - brain freeze causes a very short-lived but intense headache that may cause similar biomarker release as other headache disorders. This may be a useful human model for other headache disorders.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of one of the following: a. Diagnosis of a primary headache disorder according to the International Headache Classification, including migraine with aura, migraine without aura, chronic migraine, tension headache, cluster headache, paroxysmal hemicrania, short-lasting unilateral neuralgiform headache attacks with conjunctival injection and tearing (SUNCT), short-lasting unilateral neuralgiform headache attacks with cranial autonomic symptoms (SUNA), and hemicrania continua; b. Diagnosed by a pain medicine physician with lumbar radiculopathy (possibly including neuropathic features, nerve impingement on MRI, or electromyography (EMG) report suggestive of lumbar radiculopathy); or c. Healthy control subject with no history of debilitating headaches or debilitating back pain / radiculopathy pain, and no headaches or back pain within the previous 3 months.
* Able to provide HIPAA authorization to share prior medical records/imaging
* Age 18 and older

Exclusion Criteria:

* The following items exclude the subject from all portions of the study: a. Known history of cardiovascular or neurovascular diseases. These diseases may include carotid stenosis of >50%, vertebral stenosis, peripheral vascular disease, angina or myocardial infarction, stroke, or vascular malformations; b. History of brain tumors or epilepsy; c. Active pregnancy or lactation; d. Daily cigarette, tobacco or nicotine use; e. Life expectancy less than 1 year, co-existing disease or other characteristic that precludes appropriate diagnosis of headache or spine pain; f. Active drug / alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements; or g. Inability or unwillingness of subject to give informed consent (e.g., ward of the state)
* The following items exclude the subject only from the capsaicin portion of the study: a. Known allergy to capsaicin or hot peppers
* The following items exclude the subject only from the oxygen portion of the study: a. Pulmonary or other non-headache diseases that require the use of supplemental oxygen
* The following items exclude the subject only from the cold water irrigation (ice water) portion of the study: a. Trauma, fractures, or congenital abnormalities of the soft palate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 371 (Estimated)
Dates: Start 2018-03-21 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Activation of trigeminoautonomic reflex as assessed by change in Calcitonin gene-related peptide (CGRP) levels from before stimulation to after stimulation. | 10 minutes before pain stimulation and 10 minutes, 20 minutes, 30 minutes, 60 minutes, and 90 minutes after pain stimulation
Activation of trigeminoautonomic reflex as assessed by tear fluid production | 90 minutes after pain stimulation
  The amount of tear fluid after each intervention will be measured via Schirmer strips

SECONDARY OUTCOMES:
Activation of trigeminoautonomic reflex as assessed by change in pituitary adenylate cyclase activating polypeptide-38 (PACAP-38) levels levels from before stimulation to after stimulation. | 10 minutes before pain stimulation and 10 minutes, 20 minutes, 30 minutes, 60 minutes, and 90 minutes after pain stimulation
Activation of trigeminoautonomic reflex as assessed by saliva production | 90 minutes after pain stimulation
Activation of trigeminoautonomic reflex as assessed by nasal fluid production | 90 minutes after pain stimulation
Activation of trigeminoautonomic reflex as assessed by tactile threshold measurement with von Frey Filaments | 90 minutes after pain stimulation
Activation of trigeminoautonomic reflex as assessed by dermal blood flow | 90 minutes after pain stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Mark Burish, MD PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided